CLINICAL TRIAL: NCT04954040
Title: Clinical Trial for the Prevention and Treatment With Hydroxychloroquine + Azithromycin of Acute Respiratory Syndrome Induced by COVID-19
Brief Title: Prevention and Treatment With Hydroxychloroquine + Azithromycin of Acute Respiratory Syndrome Induced by COVID-19
Acronym: AMBUCOV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMBUCOV
Record Dates: First submitted 2021-07-06; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-04

CONDITIONS: Acute Respiratory Distress Syndrome; Covid19
Keywords: acute respiratory syndrome; SARS-CoV-2; COVID19; hydroxychloroquine; azithromycin; COVID19 symptoms
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19 | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine + Azithromycin (Experimental): Hydroxychloroquine. 1st day 200mg 2-0-2; 2nd to 5th day 200mg 1-0-1 Azithromycin. 1st day 500m 0-1-0, 2nd to 5th day 250mg 0-1-0
  Oral intake in all cases. Pills will be taken simultaneously.
  Interventions: Drug: Hydroxychloroquine Pill + Azithromycin Pill
- SOC (Standard of Care) (Active Comparator): SOC for symptoms treatment
  Acetaminophen or Metamizole, 1-1-1 Antitussives if needed
  Interventions: Drug: SOC

INTERVENTIONS:
Drug: Hydroxychloroquine Pill + Azithromycin Pill — Hydroxychloroquine. 1st day 200mg 2-0-2; 2nd to 5th day 200mg 1-0-1 Azithromycin.
  1st day 500m 0-1-0, 2nd to 5th day 250mg 0-1-0
  Arms: Hydroxychloroquine + Azithromycin
Drug: SOC — Acetaminophen or Metamizole. Antitussives if needed.
  Arms: SOC (Standard of Care)

SUMMARY:
Multi-centered, randomized, open label clinical trial to study the safety and effectivity of hydroxychloroquine + azithromycin to treat COVID-19 symptoms in primary care patients.

DETAILED DESCRIPTION:
In the patient group treated with hydroxychloroquine + azithromycin we expect to find a diminution of 20% or more regarding the evolution of acute respiratory syndrome, as opposed to patients who have not been treated with these medicines.

To date, there is no shown effective treatment regime for acute respiratory distress caused by COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patients with positive semi-quantitative PCR and COVID19 symptoms (fever, cough, diarrhea, dyspnoea, loss of smell).
* Signed informed consent

Exclusion Criteria:

* Retinal degeneration.
* Congenital or acquired long QT syndrome.
* Advanced liver failure.
* Renal insufficiency (incompatible with creatinine clearance less than 50 mL /minute).
* Allergic to hydroxychloroquine or azithromycin.
* Serious interaction with the drugs used.
* Pregnant or breastfeeding.
* Men and women in fertile and sexually active periods, who do not accept a highly effective contraceptive method.
* Inability to follow study procedures.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Hospitalization | From randomization until patient's hospitalization happens, assessed up to 28 days.
ICU admission | From date of randomization until ICU admission as a result of COVID19, assessed up to 28 days.
Death | From randomization until death by any cause related to COVID19, assessed up to 28 days.

SECONDARY OUTCOMES:
Clinical Evolution | From randomization until healing, hospitalization or death. Symptoms will be evaluated every 24 hours for a minimum of 10 days and a maximum 28 days.
  Clinical evolution will be evaluated through the following symptoms: fever, cough, dyspnoea, diarrhea, loss of smell.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Salud Priego de Córdoba, Priego de Córdoba, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after the study concludes and results are published
Supporting Information: Study Protocol, ICF, CSR
Time Frame: When study is published.
Access Criteria: Sending request.